CLINICAL TRIAL: NCT04055064
Title: Evaluating the Effects of Improving Nutritional Intake on Wound Healing in Patients With Diabetic Foot Ulcer
Brief Title: The Effects of Nutrition Supplementation and Education on the Healing of Diabetic Foot Ulcer (DFU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Raedeh Basiri, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019.26726
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Foot Ulcer
Keywords: DFU, wound healing, nutrition education,supplementation
MeSH Terms: conditions — Diabetic Foot | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): patients received nutrition education and nutritional supplements
  Interventions: Dietary Supplement: glucose control nutritional shake, nutrition education
- Control (No Intervention): patients did not receive any intervention

INTERVENTIONS:
Dietary Supplement: glucose control nutritional shake, nutrition education — Participants in the treatment group were educated about improving their diet by consuming more low-fat high-quality protein sources, vegetables, complex carbohydrates and less simple carbohydrates. They were also instructed to consume two servings (474 ml) of a commercially produced Glucose Control Nutritional Shake between meals throughout the day for 12 weeks or until complete healing. The supplements provided a total of 500 kilocalories, 28 grams of high-quality protein and essential vitamins and minerals.
  Other Names: Nutrition education
  Arms: Intervention

SUMMARY:
The overall aim of this study was to assess the effects of nutritional supplementation and education on the healing of foot ulcers in diabetic patients. The hypothesis was that improving dietary intake can promote wound healing by improving nutritional status, blood flow, and decreasing inflammatory biomarkers while increasing anti-inflammatory factors.

ELIGIBILITY:
Inclusion Criteria:

male or non-pregnant, non-lactating female ages 50 ± 20 years, diagnosis of diabetes mellitus, undergoing pharmacological treatment for glycemic control, with at least one foot with one ulcer of grade 1A based on University of Texas classification -

Exclusion Criteria:

Subjects were excluded from the study if they had HbA1c concentrations > 12%, bioengineered tissue use within four weeks prior to initial screening, a history of radiation treatment to the ulcer site, known immunosuppression, active malignancy, chronic kidney disease, liver failure/cirrhosis, heart failure and/or myocardial infarction in the past three months, use of warfarin, alcohol abuse, or any mental or physiological condition that may interfere with nutrition education and nutritional supplement intake.-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Improvement in wound healing rate(mm^2/week) | 12 weeks
  Mean change from baseline in wound area at weeks 4,8, and 12 using the following formula
  Wound Healing rate= (current area-baseline area)/time (number of weeks)
Change in inflammatory biomarkers | 12 weeks
  Mean change from baseline in c-reactive protein(ng/ml), interleukin 6(pg/ml), interleukin 10(pg/ml), and tristetraprolin(pg/ml) at weeks 4, 8, and 12
Change in lean body mass and body fat | 12 weeks
  Mean change from baseline in lean body mass(lb) and body fat(lb) at weeks 4, 8, and 12
Change in dietary intake of nutrients | 12 weeks
  Mean change from baseline in dietary intake of energy(kcal), protein(g), vitamin C(mg), vitamin E(IU), vitamin A(IU), Zinc(mg), Copper(mg), and Manganese(mg) at weeks 4, 8, and 12.

SECONDARY OUTCOMES:
Length of time that a wound achieves complete wound closure | 12 weeks
  Duration (number of days) to achieve complete wound closure from baseline assessed between both groups.
Change in basal metabolic rate | 12 weeks
  Mean change from baseline in basal metabolic rate(kcal) at weeks 4, 8, and 12.
Change in Ankle Brachial Index(ABI) | 12 weeks
  Mean change from baseline in ABI by comparing the blood pressure in the upper and lower limbs at weeks 4,8, and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
not able to share individual participant data due to IRB requirements